CLINICAL TRIAL: NCT04437394
Title: Evaluation of Functions of Swallowing and Voice in Ankylosing Spondylitis Patients
Status: Completed | Type: Observational
Sponsor: Yavuz Atar (Other)
Responsible Party: Sponsor-Investigator, Yavuz Atar, Lecturer, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: 903-19/06/2018
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Ankylosing Spondylitis; Swallowing Disorder.Other Specified; Voice Alteration
Keywords: Ankylosing spondylitis, swallowing, voice
MeSH Terms: conditions — Spondylitis, Ankylosing; Dysphonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Study group was performed on 30 patients who were diagnosed with ankylosing spondylitis using modified New York criterion.
  Interventions: Diagnostic Test: flexible endoscopic evaluation of swallowing; Diagnostic Test: The analysis of voice
- Control group: Control group was performed on 30 participants who were healthy.
  Interventions: Diagnostic Test: flexible endoscopic evaluation of swallowing; Diagnostic Test: The analysis of voice

INTERVENTIONS:
Diagnostic Test: flexible endoscopic evaluation of swallowing — The patients were assessment with flexible endoscopic swallowing evaluation was performed with colored pudding.
Diagnostic Test: The analysis of voice — Voice recordings were taken from the patients to evaluate the voice disturbance and acoustic evaluation was taken with PRAAT program.

SUMMARY:
In this study was to determine whether changes that occurred over time had an impact on the swallowing and voice functions depend of Ankylosing spondylitis patients.

DETAILED DESCRIPTION:
This study was carried out at the University of Health Sciences Okmeydani Training and Research Hospital, Department of Otorhinolaryngology. Study was performed on 30 patients and 30 healthy subjects (Group 2) who were diagnosed with ankylosing spondylitis using modified New York criterion. The patients were asked to fill the EAT-10 and flexible endoscopic swallowing evaluation was performed. Voice recordings were taken from the patients to evaluate the voice disturbance and acoustic evaluation was taken with PRAAT program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Ankylosing spondylitis
* Person who accept to consent form

Exclusion Criteria:

* Pulmoner diseases
* Laryngeal polip or nodules
* Underwent to larynx or esophageal surgery
* Central nerve system diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was performed on 30 patients who were diagnosed with ankylosing spondylitis using modified New York criterion.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Quality of swallowing | 3 months
  Quality of swallowing was assessed by Eating Assessment Tool inventory consisting in 10 questions that scores from 0 to 40. Low score is better, higher score is worse.
Values of aspiration | 3 months
  Aspiration was assessed by aspiration penetration scale during swallowing with flexible endoscopy. The scale consisting in 8 degree that scored from 1 to 8. Higher score is worse.
Voice analysis | 3 months
  Voice recordings were analyzed by PRAAT computer software. The investigator measured to shimmer, jitter and HNR voice values. The values are variation of frequency and amplitude of the sound wave. Higher value shows healthy voice for HNR parameters, lower value shows healthy voice for shimmer and jitter.
Cervical spine situation | 3 months
  Cervical spine was assessed with modify stoke ankylosing spondylitis spine score that scored from 0 to 3. Low score is better and high score is worse.
Ankylosing spondylitis disease activity | 3 months
  The investigator measured to disease activity with bath ankylosing spondylitis disease activity index consisting in 6 questions that scored from 0 to 10 and morning rigidity times. Low scores are better and high scores are worse.

SECONDARY OUTCOMES:
Demographic values | 3 months
  Demographic values were assessed as age (18-70) ,education and gender (male or female).

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Atar, Assoc. Prof., Study Director — University of Health Sciences, Istanbul Prof. Dr. Cemil Tascioglu City Hospital
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Creemers MC, Franssen MJ, van't Hof MA, Gribnau FW, van de Putte LB, van Riel PL. Assessment of outcome in ankylosing spondylitis: an extended radiographic scoring system. Ann Rheum Dis. 2005 Jan;64(1):127-9. doi: 10.1136/ard.2004.020503. Epub 2004 Mar 29. PMID 15051621
- [Result] Kelly AM, Drinnan MJ, Leslie P. Assessing penetration and aspiration: how do videofluoroscopy and fiberoptic endoscopic evaluation of swallowing compare? Laryngoscope. 2007 Oct;117(10):1723-7. doi: 10.1097/MLG.0b013e318123ee6a. PMID 17906496
- [Result] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Derived] Ahmed EA, Atar S, Atar Y, Sari H, Anarat MEA, Salturk Z, Karaketir SG, Uyar Y, Kuru O. Evaluation of the Swallowing and Voice Functions in Ankylosing Spondylitis Patients. Dysphagia. 2022 Apr;37(2):455-462. doi: 10.1007/s00455-021-10340-1. Epub 2021 Jul 14. PMID 34259915